CLINICAL TRIAL: NCT03917433
Title: Augmenting Virtual Reality Exposure Therapy for Acrophobia With Tactile Feedback and Point-based Rewards
Brief Title: Augmenting Virtual Reality Exposure Therapy for Acrophobia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: temporarily suspended recruitment due to COVID-related social distancing requirements
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Cynthia Lancaster, Assistant Professor, Clinical Psychology, University of Nevada, Reno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1345559-1
Record Dates: First submitted 2019-04-11; First posted 2019-04-17 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Specific Phobia; Anxiety Disorders; Fear of Heights; Acrophobia
Keywords: exposure therapy; virtual reality; acrophobia; fear of heights
MeSH Terms: conditions — Phobia, Specific; Anxiety Disorders; Acrophobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive virtual reality exposure therapy with tactile feedback, point-based rewards, both tactile feedback and point-based rewards, or neither tactile feedback nor point-based rewards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exposure with Tactile Feedback (Experimental): Participant completes virtual reality exposure therapy for acrophobia involving walking across a plank at higher and higher levels in a virtual city environment. In the real world, the participant walks across an actual wooden plank on the floor, which mirrors the plank in the virtual world.
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Behavioral: Tactile Feedback
- Exposure with Point-based Rewards (Experimental): Participant completes virtual reality exposure therapy for acrophobia involving walking across a plank at higher and higher levels in a virtual city environment. The participant has the opportunity to pop balloons upon reaching the ends of the plank to gain points. Participant's popping instrument in the virtual world upgrades as more points are accumulated.
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Behavioral: Point-based Rewards
- Exposure with Tactile Feedback and Point-based Rewards (Experimental): Participant completes virtual reality exposure therapy for acrophobia involving walking across a plank at higher and higher levels in a virtual city environment. In the real world, the participant walks across an actual wooden plank on the floor, which mirrors the plank in the virtual world. Also, the participant has the opportunity to pop balloons upon reaching the ends of the plank to gain points. Participant's popping instrument in the virtual world upgrades as more points are accumulated.
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Behavioral: Tactile Feedback; Behavioral: Point-based Rewards
- Virtual Reality Exposure Therapy Alone (Other): Participant completes virtual reality exposure therapy for acrophobia involving walking across a plank at higher and higher levels in a virtual city environment.
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Participant completes virtual reality exposure therapy for acrophobia involving walking across a plank at higher and higher levels in a virtual city environment.
Behavioral: Tactile Feedback — In the real world, the participant walks across an actual wooden plank on the floor, which mirrors the plank in the virtual world.
  Arms: Exposure with Tactile Feedback; Exposure with Tactile Feedback and Point-based Rewards
Behavioral: Point-based Rewards — Participant has the opportunity to pop balloons upon reaching the ends of the plank to gain points. Participant's popping instrument in the virtual world upgrades as more points are accumulated.
  Arms: Exposure with Point-based Rewards; Exposure with Tactile Feedback and Point-based Rewards

SUMMARY:
This study will examine whether tactile feedback and point-based rewards can be used to improve outcomes from virtual reality exposure therapy for acrophobia.

DETAILED DESCRIPTION:
Exposure therapy is one of the most potent techniques available for treating anxiety-related disorders, including specific phobia. However, estimates suggest that 10-48% of anxiety patients do not fully respond to exposure therapy. Meta-analyses demonstrate that virtual reality exposure therapy (VRET) is equally effective as traditional, in vivo ('in life') exposure therapy. Furthermore, individuals with anxiety disorders report greater preference (and lower likelihood of treatment refusal) for VR, rather than in vivo, exposure therapy. Although VRET has well-established efficacy and is rapidly growing in popularity, there has been very little research evaluating how specific elements of VR game design might be used to improve outcomes from VRET. This study evaluates two game design elements that we hypothesize will improve VRET outcomes: tactile feedback and a point-based reward system. Tactile feedback (TF; i.e., touching a real object that matches an element in the VR environment) enhances sense of presence in VR. Higher presence activates anxiety during VRET, which is essential for promoting the active mechanisms of exposure therapy and may also improve treatment retention. On the other hand, point-based rewards (PR) in games enhance sense of competence (i.e., sense of progress and achievement), and increase both enjoyment and likelihood of future use of games. Furthermore, several studies demonstrate that PR improves traditionally difficult-to-change health behaviors, such as increasing exercise frequency and reducing misuse of pain medications. Although this research is promising, the impact of PR on VRET is unknown. To test the influence of TF and PR on VRET outcomes, we will randomize participants with acrophobia to receive (a) standard virtual reality exposure therapy, (b) VRET with tactile feedback, (c) VRET with a point-based reward system, or (d) VRET with tactile feedback and a point-based reward system. Participants' fear reactivity will be assessed with behavioral, physiological, and subjective/self-report measures at baseline, post-treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Indicates sufficient fear of heights based on responses (a) on a self-report questionnaire (the Acrophobia Questionnaire) administered at prescreening, and (b) on Behavioral Avoidance Tests administered at baseline.

Exclusion Criteria:

* Already receiving exposure therapy for height phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral approach test (BAT)- generalization context | Change from baseline to one-month follow-up
  Participants will walk up a staircase until they reach the highest level they can complete. During each BAT, we will assess fear response behaviorally (highest step reached up to 101 steps), physiologically (heart rate and electrodermal activity), and subjectively (self reported levels of anticipated and peak fear).
Behavioral approach test (BAT) -treatment context | Change from baseline to one-month follow-up
  Participants will stand on a plank in virtual reality and raise the plank until they reach the highest level they can complete. During each BAT, we will assess fear response behaviorally (highest step reached up to 70 steps), physiologically (heart rate and electrodermal activity), and subjectively (self reported levels of anticipated and peak fear).
Acrophobia Questionnaire (AQ) | Change from baseline to one-month follow-up
  Participants will complete the AQ, a 40-item questionnaire that assesses self-reported anxiety and avoidance related to acrophobia. Scores for each subscale are summed, and totals range from 0 to 120 for each subscale, with higher scores indicating greater anxiety or avoidance.
Heights Interpretation Questionnaire (HIQ) | Change from baseline to one-month follow-up
  Participants will complete the HIQ, a 16-item questionnaire that assesses self-reported interpretations of an imagined experience of heights. Items are summed scored, and totals ranged from 16 to 80, with higher scores indicating greater height fear-relevant interpretation bias.

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule for the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 - Specific Phobia Module | Change from baseline to one-month follow-up
  Participants will be given a structured interview to determine whether they meet diagnostic criteria for specific phobia.
Treatment Drop-out Questionnaire | Post-treatment (about 1 week)
  Experimenters will record whether or not participants drop out of treatment. This will be operationalized as beginning virtual reality exposure therapy, but discontinuing the study before the two-session treatment is complete.
Willingness to continue exposure therapy | Post-treatment (about 1 week)
  This scale will assess assess whether participants would be willing (from 0% to 100%) to use the heights exposure program at home, or to return to the lab for another therapy session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
Study protocols and de-identified data will be shared at the request of other researchers.